CLINICAL TRIAL: NCT00970957
Title: Study of the Safety and Efficacy of Bevacizumab Intravitreal Injections for the Treatment of Macular Edema Secondary to Retinal Vein Occlusions
Brief Title: Safety and Effectiveness of Bevacizumab Intravitreal Injections in the Treatment of Macular Edema Secondary to Retinal Vein Occlusion
Acronym: EBOVER
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Instituto Universitario de Oftalmobiología Aplicada (Institute of Applied Ophthalmobiology) - IOBA (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IOBA-03-2008; EUDRA -CT 2008-005789-30
Record Dates: First submitted 2009-09-02; First posted 2009-09-03 (Estimated); Last update posted 2014-03-19 (Estimated); Status verified 2014-03

CONDITIONS: Macular Edema; Retinal Vein Occlusion
Keywords: Macular edema; Retinal Vein Occlusion; Bevacizumab
MeSH Terms: conditions — Macular Edema; Retinal Vein Occlusion | interventions — Bevacizumab; salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor

ARMS (4):
- Central RVO - Macular edema - Avastin (Experimental): Patients with Macular edema secondary to CENTRAL Retinal Vein Occlusion that will be treated with intravitreal injection of avastin once per month during the first 3 months. Re-treatments will be given as per protocol.
  Interventions: Drug: Avastin Intravitreal Injection
- Central RVO - Macular edema - Sham (Sham Comparator): Patients with Macular edema secondary to CENTRAL Retinal Vein Occlusion that will have a sham procedure performed. Injection without needle.
  Interventions: Drug: Sham Avastin Intravitreal Injection
- Branch RVO - Macular edema - Avastin (Experimental): Patients with Macular edema secondary to BRANCH Retinal Vein Occlusion that will be treated with intravitreal injection of avastin once per month during the first 3 months. Re-treatments will be given as per protocol.
  Interventions: Drug: Avastin Intravitreal Injection
- Branch RVO - Macular edema - Sham (Sham Comparator): Patients with Macular edema secondary to BRANCH Retinal Vein Occlusion that will have a sham procedure performed. Injection without needle.
  Interventions: Drug: Sham Avastin Intravitreal Injection

INTERVENTIONS:
Drug: Avastin Intravitreal Injection — Intravitreal injection of 1.25mg Avastin (Bevacizumab) per month, during the first 3 months. Retreatments will be required if visual acuity or macular edema thickness worsen as defined per protocol
  Other Names: Avastin
  Arms: Branch RVO - Macular edema - Avastin; Central RVO - Macular edema - Avastin
Drug: Sham Avastin Intravitreal Injection — Intravitreal Injection simulation with a syringe without needle. The rest of the procedure remains the same as if intravitreal injection were to be performed (antibiotic prophylaxis, local anesthesia, ...).
  Other Names: Sham
  Arms: Branch RVO - Macular edema - Sham; Central RVO - Macular edema - Sham

SUMMARY:
Lack of an effective treatment for macular edema secondary to central retinal vein occlusion and the bad response to grid laser treatment in patients with macular edema secondary to branch retinal vein occlusion, together with the high incidence of the pathology and the great functional loss in the patients that suffer from it has motivated the search for new therapeutic approaches.

In recent times, intravitreal bevacizumab has been tested in clinical practice in small series of patients with this pathology, whether as first treatment or after failure of grid laser treatment with good functional results in short series.

However, no retreatment information is available, although preliminary results from published series are good.

ELIGIBILITY:
Inclusion Criteria:

* Patient male or female 18 years old or more
* Foveal macular edema secondary to Retinal Vein Occlusion confirmed by Fluorescein angiography and Optical Coherence Tomography, with a subcentral field thickness of at least 250 microns
* Patients with best corrected visual acuity loss within the last 6 months of evolution, caused by the macular edema as stated by investigator´s judgement.
* Best corrected visual acuity tested by ETDRS within 20/40 and 20/400 in the study eye.
* Signed Informed consent.
* Signed Data Protection Consent.
* Negative pregnancy test before entering the study for childbearing potential women, who must commit to use a medically accepted contraceptive method for the whole study.
* Macular Subcentral field assessed by Ocular coherence tomography of at least 250 microns thick.
* No presence of eye opacities that may prevent fundus exploration. No condition that may prevent correct eye dilation.
* No known allergy to fluorescein.
* Only an eye per patient will be included in the study,even if both eyes have the pathology.

Exclusion Criteria:

* Macular edema secondary to any other condition such as: diabetes retinopathy, hypertension, Juxtafoveal telangiectasia, ...
* Any previous treatment for macular edema such as photocoagulation, vitrectomy, triamcinolone, radial optic neurotomy, ... in the study eye.
* Any ocular illness thay may be associated to increased/high levels of VEGF (Age related macular degeneration, Diabetes retinopathy, Uveitis, ...)
* Systemical illnesses thay may be associated to increased/high levels of VEGF (e.g. tumours).
* Medical history of brain vascular episodes (stroke), ictus, angor pectoris or myocardial infarct within 3 months before study inclusion.
* Pregnancy or nursing.
* Hypersensibility known or suspected to Bevacizumab, his excipients or any related molecule.
* Uncontrolled hypertension refractary to medical treatment.
* Participation in any other trial or study within the last 3 months (minerals and vitamins excluded) or treatment with anti-VEGF in the non-study eye within the previous 3 months.
* Tractional maculopathy and/or epiretinal membrane assessed by Ocular Coherence Tomography.
* Media opacities that don´t allow correct eye exploration and fundus examination/photographs.
* Cataract surgery / Yag capsulotomy within the previous 6 months.
* Filtration surgery.
* Previous medical history of ocular illnesses as: viral infections, inflammatory pathology, serous central choroidopathy, retinal detachment or any other illness that may have an influence in visual acuity.
* Presence of foveal atrophy, severe pigmentary changes, dense subfoveal haemorrhages, confluent subfoveal hard exudates or any other condition that may influence functional recovery of the macular edema.
* Cataract that may be responsible for additional visual acuity loss of more than 2/10.
* Medically uncontrolled intraocular pressure higher than 25 mm Hg.
* External ocular illnesses active at inclusion as: conjunctivitis, blepharitis, eye sore, ...

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2009-09; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Best corrected visual acuity assessed as described in the Early Treatment for Diabetes Retinopathy Study (ETDRS) | 1 month

SECONDARY OUTCOMES:
Macular Subcentral Field Thickness assessed by Ocular coherence tomography | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: María Isabel López Gálvez, MD, PhD, Principal Investigator — IOBA - Instituto Universitario de Oftalmobiología Aplicada
Locations (13):
- Spain (13):
  - Instituto Oftalmológico de Alicante, Alicante, Alicante
  - Hospital de la Vall D´Hebrón, Barcelona, Barcelona
  - Hospital Clinic, Barcelona, Barcelona
  - Hospital Provincial Conxo - Fundación IDICHUS, Santiago de Compostela, La Coruña
  - Hospital Clínico San Carlos, Madrid, Madrid
  - Hospital Ramón y Cajal, Madrid, Madrid
  - Hospital La Paz, Madrid, Madrid
  - Hospital General Reina Sofía, Espinardo, Murcia
  - Clínica Universitaria de Navarra, Pamplona, Navarre
  - Hospital Virgen de la Macarena, Seville, Sevilla
  - Hospital Virgen de Valme, Seville, Sevilla
  - Hospital General Universitario de Valencia, Valencia, Valencia
  - Instituto Universitario de Oftalmobiología Aplicada, Valladolid, Valladolid